CLINICAL TRIAL: NCT03508908
Title: Impact of a Novel HIV-1 RNA Testing Intervention to Detect Acute and Prevalent HIV Infection and Reduce HIV Transmission - Tambua Mapema Plus
Brief Title: Tambua Mapema Plus - to Discover HIV Infection Early and Prevent Onward Transmission
Acronym: TMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Washington (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, DrEduard Sanders, Public Health Physician and Epidemiologist, University of Oxford
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: DAIDS-ES ID 38181; 1R01AI124968-01A1 (NIH)
Record Dates: First submitted 2018-03-07; First posted 2018-04-26 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections
Keywords: HIV testing; ART; partner notification; PrEP
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: This trial will use a modified stepped wedge design to evaluate the yield of the HIV-1 RNA testing intervention at 6 public or private health facilities in Kenya, before (1,375 patients) and after (1,500 patients) intervention delivery. This study will be conducted in two phases (observation phase and intervention phase) at each site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Observation Period (No Intervention): HIV testing will only be done if ordered by the primary care clinician. Individuals diagnosed with HIV who have not yet notified partners will be offered assisted partner notification at a 6-week visit.
- Intervention Period (Active Comparator): Combination intervention with HIV-1 RNA testing followed by rapid tests if positive for HIV diagnosis, immediate ART if diagnosed, assisted partner notification with HIV-1 RNA testing of partners, and PrEP for uninfected partners in discordant relationships.
  Interventions: Diagnostic Test: HIV-1 RNA testing

INTERVENTIONS:
Diagnostic Test: HIV-1 RNA testing — During the intervention period, a blood sample will be obtained and tested for AHI using point-of-care Xpert® HIV Qual assay (Cepheid, Sunnyvale, California, USA). Individuals who test positive will undergo rapid tests to differentiate acute from prevalent HIV infection. Newly diagnosed individuals will be offered immediate ART and assisted partner notification with the HIV-1 RNA testing intervention delivered to partners following the same approach.
  Other Names: Xpert HIV-1 RNA testing
  Arms: Intervention Period

SUMMARY:
This study will assess the impact of an HIV-1 RNA testing intervention targeting adult patients aged 18-39 years who seek urgent care for symptoms at primary care facilities and meet specific risk criteria for acute HIV infection. All newly diagnosed HIV-infected patients in the intervention arm will be linked to care and offered both immediate treatment and assisted partner notification. Partners will also be tested using the HIV testing intervention, and pre-exposure prophylaxis will be offered to uninfected individuals with HIV-infected partners. The cost-effectiveness of this intervention will be evaluated.

DETAILED DESCRIPTION:
This is a proof-of-concept study comparing outcomes of a health facility-based acute HIV infection (AHI) and prevalent HIV testing intervention using point of care HIV-1 RNA detection, combined with assisted partner services (aPS) and follow-up in an antiretroviral therapy (ART) cohort for all newly diagnosed individuals and follow-up in a pre-exposure prophylaxis (PrEP) cohort for the uninfected partners of newly diagnosed individuals, compared to standard care.

Study Design: Randomized stepped-wedge study with prospective cohort follow-up of all individuals newly diagnosed with acute or prevalent HIV infection and of up to 300 identified partners of these persons. Individuals enrolled in the observation phase will be compared to those enrolled in the intervention phase at each facility, after undergoing the following procedures in each phase.

Study Population: The study population will be recruited from among male and female adult patients who present for care at 6 public or private outpatient clinics in coastal Kenya. Eligibility criteria for the HIV-1 RNA testing intervention include: 1) age from 18-39 years; 2) not previously diagnosed with HIV infection; and 3) a score ≥2 on our AHI risk score algorithm. Eligibility criteria for partners of newly diagnosed cases with acute or prevalent HIV infection include: 1) age over 18 years; and 2) not previously diagnosed with HIV infection.

Sample Size: 3,175 study participants total, including 2,875 participants in the stepped-wedge study (1,375 in the observation period and 1,500 in the intervention period). We estimate that approximately 2% of participants in the observation period (n=28) and approximately 5% of participants in the intervention period (n=75) will test positive for HIV infection and continue in the study. We estimate that up to 300 partners of newly diagnosed individuals will be offered enrollment and tested for HIV using standard tests (observation period) or HIV-1 RNA testing (intervention period).

Participating Sites: Kenya Medical Research Institute (KEMRI)-Wellcome Trust Programme, Kilifi, Kenya with stepped wedge trial implementation at 6 community health facilities (2-4 public, 2-4 private) and ART and PrEP cohort follow-up at the KEMRI Research Clinic in Mtwapa, Kenya.

Schedule of Procedures: Individuals eligible for the HIV-1 RNA testing intervention will be offered enrollment when they seek care at one of the study facilities, with testing taking place on that same day. For individuals with negative test results for both acute and prevalent HIV infection, no further follow-up will occur. One 6-week follow-up visit will occur after testing for all individuals who are newly diagnosed with HIV. Procedures for the aPS intervention, the ART cohort, and the PrEP cohort are detailed in this protocol.

Study Duration: Study enrollment will occur over 24 months. Following enrollment and study procedures (1-2 hours of time), all participants who test negative for HIV infection will have no further visits. All participants newly diagnosed with HIV will have a 6-week follow-up visit. All participants who enroll in the ART or PrEP cohort will be followed for a total of 12 months.

Intervention: Testing for acute and prevalent HIV infection, followed by partner notification services and immediate ART (provided by the Kenyan Ministry of Health) for newly diagnosed individuals and PrEP (provided by Gilead) for uninfected partners in serodiscordant relationships.

ELIGIBILITY:
Inclusion Criteria:

* age from 18-39 years;
* not previously diagnosed with HIV infection; and
* a score ≥2 on our risk score algorithm to identify persons at higher risk for AHI, with scoring as follows:

  * age 18-29 years (1),
  * fever (1),
  * fatigue (1),
  * body pains (1),
  * diarrhea (1),
  * sore throat (1), and
  * genital ulcer disease (GUD) (3).

Eligibility criteria for partners of newly diagnosed cases with prevalent or acute HIV include:

* age over 18 years; and
* not previously diagnosed HIV infection.

Exclusion Criteria:

Patients not meeting inclusion criteria or those who are not willing or able to participate (e.g., due to illness or time constraints, or at the discretion of the study clinician) will be excluded.

Individuals at high risk for Intimate Partner Violence (IPV) are excluded from the aPS intervention, but eligible for all other components of the study.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2887 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SUSAN M GRAHAM, MD MPH PHD, Principal Investigator — University of Washington; EDUARD J SANDERS, MD MPH PHD, Principal Investigator — University of Oxford
Locations (1):
- KEMRI Mtwapa, Kilifi, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Babigumira JB, Agutu CA, Hamilton DT, van der Elst E, Hassan A, Gichuru E, Mugo PM, Farquhar C, Ndung'u T, Sirengo M, Chege W, Goodreau SM, Sanders EJ, M Graham S. Testing strategies to detect acute and prevalent HIV infection in adult outpatients seeking healthcare for symptoms compatible with acute HIV infection in Kenya: a cost-effectiveness analysis. BMJ Open. 2022 Sep 29;12(9):e058636. doi: 10.1136/bmjopen-2021-058636. PMID 36175097
- [Derived] Agutu CA, Oduor TH, Hassan AS, Mugo PM, Chege W, de Wit TFR, Sanders EJ, Graham SM. Predictors of testing history and new HIV diagnosis among adult outpatients seeking care for symptoms of acute HIV infection in coastal Kenya: a cross-sectional analysis of intervention participants in a stepped-wedge HIV testing trial. BMC Public Health. 2022 Feb 11;22(1):280. doi: 10.1186/s12889-022-12711-1. PMID 35148720
- [Derived] Sanders EJ, Agutu C, van der Elst E, Hassan A, Gichuru E, Mugo P, Farquhar C, Babigumira JB, Goodreau SM, Hamilton DT, Ndung'u T, Sirengo M, Chege W, Graham SM. Effect of an opt-out point-of-care HIV-1 nucleic acid testing intervention to detect acute and prevalent HIV infection in symptomatic adult outpatients and reduce HIV transmission in Kenya: a randomized controlled trial. HIV Med. 2022 Jan;23(1):16-28. doi: 10.1111/hiv.13157. Epub 2021 Aug 25. PMID 34431196
- [Derived] Graham SM, Agutu C, van der Elst E, Hassan AS, Gichuru E, Mugo PM, Farquhar C, Babigumira JB, Goodreau SM, Hamilton DT, Ndung'u T, Sirengo M, Chege W, Sanders EJ. A Novel HIV-1 RNA Testing Intervention to Detect Acute and Prevalent HIV Infection in Young Adults and Reduce HIV Transmission in Kenya: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Aug 7;9(8):e16198. doi: 10.2196/16198. PMID 32763882

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We identified the participating health facilities (three in Kilifi county; three in Mombasa county) due to their size, location (within 20 km of our KEMRI Research Clinic), patient volume (> 500 patients aged 18-39 years seen over 3 months) and willingness to collaborate with the research team. All clinics served general population patients; the four public facilities included offered limited programming for key populations. Some sites had minor delays in starting an intervention period.
Pre-assignment Details: We used a modified stepped-wedge design to evaluate outcomes before and after intervention delivery. Six clinics each had two phases (observation and intervention), for 12 clinic periods. Each clinic period lasted 6 months or until 250 participants were recruited, except first clinic period (3 months of observation, 125 participants). The order in which clinics were active was randomized such that only 2 clinics provided the intervention at a given time (due to limited testing platforms).
Units Other Than Participants: Clinic periods
Groups:
- Observation Period: During the observation period, clinics provided standard care, and participants were enrolled, completed a standardized tablet-based survey, and followed up to determine whether the clinic staff provided HIV testing at the index visit.
- Intervention Period: During the intervention period, all participants enrolled were offered opt-out HIV testing using the HIV-1 NAAT intervention. In addition, participants completed the same standard tablet-based survey as in the observation period.
- Observation Period Partners: Partners identified in the observation period who had not been tested by 6 weeks were offered testing as part of the research study.
- Intervention Period Partners: Partners identified in the intervention period were offered enhanced HIV testing as part of the intervention.
Period: Month 0-3
Arm/Group | Observation Period | Intervention Period | Observation Period Partners | Intervention Period Partners
Started | 249; 2 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods
Completed | 249; 2 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods
Not Completed | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods
Period: Month 4-6
Arm/Group | Observation Period | Intervention Period | Observation Period Partners | Intervention Period Partners
Started | 250; 2 Clinic periods | 125; 1 Clinic periods | 1; 1 Clinic periods | 1; 1 Clinic periods
Completed | 250; 2 Clinic periods | 125; 1 Clinic periods | 1; 1 Clinic periods | 1; 1 Clinic periods
Not Completed | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods
Period: Month 7-9
Arm/Group | Observation Period | Intervention Period | Observation Period Partners | Intervention Period Partners
Started | 250; 2 Clinic periods | 250; 2 Clinic periods | 1; 1 Clinic periods | 1; 1 Clinic periods
Completed | 250; 2 Clinic periods | 250; 2 Clinic periods | 1; 1 Clinic periods | 1; 1 Clinic periods
Not Completed | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods
Period: Month 10-12
Arm/Group | Observation Period | Intervention Period | Observation Period Partners | Intervention Period Partners
Started | 250; 2 Clinic periods | 250; 2 Clinic periods | 0; 0 Clinic periods | 2; 2 Clinic periods
Completed | 250; 2 Clinic periods | 250; 2 Clinic periods | 0; 0 Clinic periods | 2; 2 Clinic periods
Not Completed | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods
Period: Month 13-15
Arm/Group | Observation Period | Intervention Period | Observation Period Partners | Intervention Period Partners
Started | 250; 2 Clinic periods | 250; 2 Clinic periods | 0; 0 Clinic periods | 2; 2 Clinic periods
Completed | 250; 2 Clinic periods | 250; 2 Clinic periods | 0; 0 Clinic periods | 2; 2 Clinic periods
Not Completed | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods
Period: Month 16-18
Arm/Group | Observation Period | Intervention Period | Observation Period Partners | Intervention Period Partners
Started | 125; 1 Clinic periods | 250; 2 Clinic periods | 1; 1 Clinic periods | 1; 1 Clinic periods
Completed | 125; 1 Clinic periods | 250; 2 Clinic periods | 1; 1 Clinic periods | 1; 1 Clinic periods
Not Completed | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods
Period: Month 19-21
Arm/Group | Observation Period | Intervention Period | Observation Period Partners | Intervention Period Partners
Started | 0; 0 Clinic periods | 250; 2 Clinic periods | 0; 0 Clinic periods | 3; 2 Clinic periods
Completed | 0; 0 Clinic periods | 250; 2 Clinic periods | 0; 0 Clinic periods | 3; 2 Clinic periods
Not Completed | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods
Period: Month 22-24
Arm/Group | Observation Period | Intervention Period | Observation Period Partners | Intervention Period Partners
Started | 0; 0 Clinic periods | 125; 1 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods
Completed | 0; 0 Clinic periods | 125; 1 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods
Not Completed | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods | 0; 0 Clinic periods

BASELINE CHARACTERISTICS:
Population: Overall, we enrolled 1374 participants during the observation period and 1500 participants during the intervention period. Thirteen partners of index patients newly diagnosed with HIV consented for HIV testing within the study: 3 in the observation period and 10 in the intervention period.
Groups:
- Observation Period Partners: Consented for testing at week 6
- Intervention Period Partners: Consented for testing and follow-up as soon as possible after diagnosis of the index patient
- Total: Total of all reporting groups
Arm/Group | Observation Period | Intervention Period | Observation Period Partners | Intervention Period Partners | Total
Number analyzed (Participants) | 1374 | 1500 | 3 | 10 | 2887
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Age was missing for 6 partners in the intervention period.
  years | 25 [23 to 29] | 26 [23 to 30] | 32.6 [28.2 to 35.8] | 32.4 [28.7 to 34.6] | 25 [23 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 886 | 887 | 2 | 3 | 1778
  Male | 488 | 613 | 1 | 7 | 1109
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1374 | 1500 | 3 | 10 | 2887
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 1374 | 1500 | 3 | 10 | 2887
HIV testing history [Count of Participants; unit: Participants] — Population: HIV testing history was missing for 7 partners in the intervention period.
  Participants
    Never tested for HIV | 147 | 153 | 1 | 2 | 303
    Tested for HIV in past 12 months | 499 | 563 | 1 | 1 | 1064
    Tested for HIV over 12 months ago | 728 | 784 | 1 | 0 | 1513
    Missing | 0 | 0 | 0 | 7 | 7

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Newly Diagnosed HIV Infection at Care Seeking
Description: Primary endpoints for the HIV-1 RNA testing intervention include the proportion of participants with newly diagnosed prevalent or AHI at care seeking.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Adult Outpatients With Symptoms of Acute HIV Infection: Adult symptomatic outpatients aged 18-39 years were evaluated by a consensus AHI risk score. Patients with a risk score ≥2 and no previous HIV diagnosis were enrolled in a stepped-wedge trial of opt-out delivery of point-of-care (POC) HIV-1 nucleic acid testing (NAAT), compared to standard provider-initiated HIV testing using rapid tests in the observation period.
- Observation Phase; Intervention Phase: adult participants aged 18-39 years
Arm/Group | Adult Outpatients With Symptoms of Acute HIV Infection | Observation Phase | Intervention Phase
Number analyzed (Participants) | 2874 | 1374 | 1500
Participants
  HIV-positive | 50 | 13 | 37
  Acute HIV infection | 2 | 0 | 2
  HIV-negative | 2822 | 1361 | 1461

2. Secondary Outcome: Proportion of Newly Diagnosed Patients Linked to Care
Description: Secondary endpoints for the linkage to care intervention include the proportion of newly diagnosed patients captured in the HIV care cascade.
Time Frame: 24 months
Population: newly diagnosed participants
Measure: Count of Participants; unit: Participants
Arm/Group | Observation Period | Intervention Period
Number analyzed (Participants) | 13 | 37
Participants | 9 | 33

3. Secondary Outcome: Proportion of Named Partners Tested for HIV
Description: Proportion of named partners tested for HIV in each period
Time Frame: 24 months
Population: In each period, trial participants who were newly diagnosed with HIV infection were offered assisted partner notification services and asked to report partners. Named partners who were successfully contacted were offered HIV testing and, if willing, provided informed consent for testing and documentation of the test result as part of this trial. Not all named partners were consented. Tested partners were referred to an observational HIV or PrEP cohort according to their status.
Measure: Count of Participants; unit: Participants
Groups:
- Observation Period: Observation period index participants who were newly diagnosed with HIV were asked about partner outcomes 6 weeks after diagnosis.
- Intervention Period: Intervention period index participants who were newly diagnosed with HIV were offered assisted partner notification services and partners were assessed by the study team 6 weeks after diagnosis.
Arm/Group | Observation Period | Intervention Period
Number analyzed (Participants) | 15 | 66
Participants | 3 | 10

4. Secondary Outcome: Cost Effectiveness of Novel RNA Testing Intervention: Total Cost (Including Both Testing and HIV-positive Patient Management) Per Participant (Base Case Patient Modeled)
Description: Model outputs will include an analysis of the cost effectiveness of the novel testing intervention assessing several parameters of the HIV prevention and care cascade using stochastic, agent-based mathematical modelling. The population of interest modeled was 18- to 39-year-old heterosexuals in Kenya. The age range coincides with the sampled population in this study (NCT03508908) which provided the majority of the parameters for the networks and behavioral modules in the simulation. The observations from this study were weighted to match the sex and age composition reported in the Kenya Fact and Figures 2015 published by the Kenya National Bureau of Statistics. Additional model parameters were drawn from the literature on HIV infection, prevention, and treatment in Kenya.The analysis was conducted over a time horizon of 10 years, consistent with the mathematical model. 10,000 base-case patients (simulations) were run.
Time Frame: Data collected over 2 years, data is a predicted time point extrapolated to 10 years
Population: The total cost (including both testing and HIV-positive patient management) per participant(base case patient modeled) is derived from the model where a measure of dispersion was not an output of the model.
Measure: Number; unit: US dollars
Units Other Than Participants: case simulations
Groups:
- Observation Phase: The population of interest modeled was 18- to 39-year-old heterosexuals in Kenya.The age range coincides with the sampled population in this study (NCT03508908) which provided the majority of the parameters for the networks and behavioral modules in the simulation. The observations from this study were weighted to match the sex and age composition reported in the Kenya Fact and Figures 2015published by the Kenya National Bureau of Statistics.
- Intervention Phase: The population of interest modeled was 18- to 39-year-old heterosexuals in Kenya.The age range coincides with the sampled population in this study (NCT03508908) which provided the majority of the parameters for the networks and behavioral modules in the simulation. The observations from this study were weighted to match the sex and age composition reported in the Kenya Fact and Figures 2015 published by the Kenya National Bureau of Statistics.
Arm/Group | Observation Phase | Intervention Phase
Number analyzed (Participants) | 1374 | 1500
Number analyzed (case simulations) | 10000 | 10000
US dollars | 47.24 | 214.91

5. Secondary Outcome: Cost Effectiveness of Novel RNA Testing Intervention: Disability-Adjusted Life Years (Base Case Patient Modeled)
Description: Disability-adjusted Life Year (DALY) is an index calculated as the sum of years of life lost (YLL) plus the years lost due to disability (YLD), where 1 DALY represents one lost year of healthy life. The higher the DALY index value, the worse the outcome, where there is no theoretical minimum ore maximum index value. the sampled population in this study (NCT03508908) which provided the majority of the parameters for the networks and behavioral modules in the simulation. The observations from this study were weighted to match the sex and age composition reported in the Kenya Fact and Figures 2015 published by the Kenya National Bureau of Statistics. Additional model parameters were drawn from the literature on HIV infection, prevention, and treatment in Kenya. The analysis was conducted over a time horizon of 10 years, consistent with the mathematical model. 10,000 base-case patients (simulations) were run.
Time Frame: Data collected over 2 years, data is a predicted time point extrapolated to 10years
Measure: Number; unit: index
Units Other Than Participants: case simulations
Arm/Group | Observation Phase | Intervention Phase
Number analyzed (Participants) | 1374 | 1500
Number analyzed (case simulations) | 10000 | 10000
index | 0.2140 | 0.1598
Statistical Analysis 1: Comparison: Observation Phase vs Intervention Phase; Cost (in US dollars) per DALY averted (Intervention referenced to Observation); Test type: Other; US dollars per DALY averted = 3098 — Cost (in US dollars) per DALY averted (Intervention referenced to Observation)

ADVERSE EVENTS:
Time Frame: Adverse events for those tested at a single clinic visit but not diagnosed with HIV were evaluated on that same day. Adverse events for those diagnosed with HIV were evaluated over the subsequent 6 weeks. Adverse events for those in cohort follow-up were evaluated over the entire 12-month follow-up period.
Description: We evaluated for social harms of the HIV testing and partner notification services components of the intervention, with a focus on intimate partner violence.
Groups:
- Intervention Period Partners: Partners of intervention period index patients were offered HIV testing and consented if willing.
Arm/Group | Observation Period | Intervention Period | Observation Period Partners | Intervention Period Partners
All-Cause Mortality (participants affected / at risk) | 0/1374 | 0/1500 | 0/3 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/1374 | 0/1500 | 0/3 | 0/10
Other Adverse Events (participants affected / at risk) | 0/1374 | 0/1500 | 0/3 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT03508908/Prot_SAP_ICF_002.pdf